CLINICAL TRIAL: NCT05598073
Title: Racial Differences in Yoga-Induced Cardiovascular and Immune Responses
Brief Title: Racial Differences in Yoga-Induced Responses
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The student leading the project decided not to continue.
Sponsor: Texas State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 6877
Record Dates: First submitted 2020-01-08; First posted 2022-10-28 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2020-01

CONDITIONS: Cardiovascular and Immune Responses to Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1-hour vinyasa yoga session (Experimental): Participants will complete a 1-hour vinyasa yoga DVD.
  Interventions: Behavioral: Vinyasa yoga session

INTERVENTIONS:
Behavioral: Vinyasa yoga session — One hour of vinyasa yoga will be completed.

SUMMARY:
The purpose of this study is to 1) determine whether racial differences are evident in resting arterial stiffness and ambulatory blood pressure between African Americans and Caucasians 2) compare heart rate, blood pressure and cytokine production responses to exercise (yoga) between African Americans and Caucasians; 3) compare isokinetic muscular strength between racial groups; and 4) determine if correlations exist between these measures.

ELIGIBILITY:
Inclusion Criteria:

* Men between the ages of 18 and 39 (25 African American and 25 Caucasian) that are not professional or collegiate athletes
* Must exercise at least 3 days per week and have no more than 1 month of yoga practice.

Exclusion Criteria:

* Having stage 2 hypertension (>130 mmHg for systolic / >90 mmHg for diastolic) or higher or having taken BP medications within the 3 months prior to testing
* Infection within the previous 4 weeks
* Known renal disease
* Prior myocardial infarction
* Known coronary artery disease
* Personal history of stroke
* Heart failure
* Cardiac arrhythmias
* Chronic obstructive pulmonary disease
* Recent chest pain or dyspnea
* Orthopedic limitations that preclude the execution of yoga postures
* Current insulin dependence
* Chronic inflammatory conditions
* Blindness or deafness as participants will need to follow a yoga DVD in order to complete the session
* Having practiced yoga for more than 1 month
* Having parents of mixed racial backgrounds (i.e. both parents must be Caucasian or African American)
* Not being African American or Caucasian
* Being a professional or collegiate athlete
* Being insulin-dependent

Ages: 18 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-15 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Arterial stiffness | Once at baseline
  Cardio-ankle vascular index
Ambulatory blood pressure | Once at baseline
  24 hours of ambulatory blood pressure monitoring
Isokinetic strength | Once at baseline
  Isokinetic leg extension and flexion strength assessments at 60,120,210,300, and 400 degrees per second
Inflammatory markers | Once at baseline
  Blood samples will be obtained and analyzed for interleukin-6 and tumor necrosis factor alpha
Inflammatory markers | Once 30 minutes into the 1-hour yoga session
  Blood samples will be obtained and analyzed for interleukin-6 and tumor necrosis factor alpha
Inflammatory markers | Once immediately after the 1-hour yoga session
  Blood samples will be obtained and analyzed for interleukin-6 and tumor necrosis factor alpha

CONTACTS AND LOCATIONS:
Locations (1):
- Stacy Hunter, San Marcos, Texas, United States

IPD SHARING:
Plan to Share IPD: No